CLINICAL TRIAL: NCT00712322
Title: A 14-day, Open-label, Multicenter, Dose-escalating, Sequential Cohort Study to Evaluate Pharmacodynamics (Urodynamics) and Pharmacokinetics, Clinical Efficacy, Tolerability and Safety Following Multiple Doses (mg/kg/Day) of a Darifenacin Liquid Oral Suspension Given BID in Children, Ages 2 - 15 Years, With Neurogenic Detrusor Overactivity
Brief Title: A Two-week Open-label Pharmacodynamic and Pharmacokinetic Study of Multiple Doses of a Darifenacin Liquid Oral Suspension in Children (2 - 15 Years) With Neurogenic Detrusor Overactivity
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to extremely difficult enrollment.
Sponsor: Warner Chilcott (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CDAR328B2201
Record Dates: First submitted 2008-07-03; First posted 2008-07-09 (Estimated); Results first posted 2022-06-09 (Actual); Last update posted 2022-06-09 (Actual); Status verified 2021-09

CONDITIONS: Neurogenic Detrusor Overactivity
Keywords: Pediatric, Children, Urodynamics, Oral Suspension, Overactive bladder, Dose-finding, Neurogenic Detrusor Overactivity, Meningomyelocele, Spinal cord injury
MeSH Terms: conditions — Urinary Bladder, Overactive; Meningomyelocele; Spinal Cord Injuries | interventions — darifenacin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort 1 (Darifenacin 0.030 mg/kg/day) (Experimental): Following a 7-day washout period, participants received darifenacin liquid oral suspension, 0.030 milligrams/kilogram/day (mg/kg/day) dispensed per twice a day (BID) dosing, for 14 days.
  Interventions: Drug: Darifenacin
- Cohort 2 (Darifenacin 0.0625 mg/kg/day) (Experimental): Following a 7-day washout period, participants received darifenacin liquid oral suspension, 0.0625 mg/kg/day dispensed per BID dosing, for 14 days.
  Interventions: Drug: Darifenacin
- Cohort 3 (Darifenacin 0.125 mg/kg/day) (Experimental): Following a 7-day washout period, participants received darifenacin liquid oral suspension, 0.125 mg/kg/day dispensed per BID dosing, for 14 days.
  Interventions: Drug: Darifenacin

INTERVENTIONS:
Drug: Darifenacin — Following a 7-day washout period, participants received darifenacin liquid oral suspension up to 14 days.
  Other Names: Enablex®, Emselex®, DAR328

SUMMARY:
This study will evaluate the pharmacodynamics and pharmacokinetics of darifenacin liquid oral suspension in children, ages 2-15 years, with neurogenic detrusor overactivity. The results will support a benefit-risk based dosage recommendation for phase IIIa clinical trials.

ELIGIBILITY:
Inclusion Criteria:

* Male and female participants ages 2-15 years
* Documented detrusor overactivity associated with a known neurological condition such as meningomyelocele or spinal cord injury, and confirmed by urodynamics at baseline
* Using clean intermittent catheterization (CIC) on a regular basis
* Participating in a bowel program on a regular basis
* Able to swallow the study medication in accordance to the protocol
* Participants and/or parent/guardian able to complete the bladder diary and follow the study procedures

Exclusion Criteria:

* Treatment with drugs known to significantly affect the urinary bladder and urinary bladder outlet function
* Fecal impaction. Participants may be included, once this condition has resolved
* Clinically significant anatomical abnormalities or acquired disorders of the urinary tract
* Previous reconstructive surgery (augmentation etc.) of the bladder or bladder outlet
* Symptomatic urinary tract infection unresolved at time of urodynamic study and/or completion of bladder diary.
* Diabetes insipidus
* Electro stimulation therapy or bladder training within 2 weeks prior to Visit 1 and at any time during the study
* Concomitant diseases, in which the use of darifenacin is contraindicated
* History of hypersensitivity to darifenacin or to drugs with similar chemical structures
* Participants with any physical and cognitive impairment or any other condition which in the opinion of the investigator makes the participants unsuitable for inclusion
* Female adolescent of child-bearing potential, unless using an acceptable method of contraception
* Pregnant or nursing (lactating) female adolescents Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 2 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 35 (Actual)
Dates: Start 2008-10-07 (Actual); Primary Completion 2013-05-23 (Actual); Study Completion 2013-05-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Herman Ellman, MD, Study Director — Warner Chilcott (US) LLC
Locations (12):
- United States (9):
  - University of California at San Diego, San Diego, California
  - Children's Hospital, Karp 8210, Boston, Massachusetts
  - Children's Hospital of Michigan, Detroit, Michigan
  - Washington University Pediatric Urology, St Louis, Missouri
  - Pediatric Urology Associates, PC, Lake Success, New York
  - Pediatric Urology Associates PC, Tarrytown, New York
  - Pediatric & Adolescent Urology, Inc Akron Children's Hospital, Akron, Ohio
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Oregon Health & Science University, Portland, Oregon
- Colombia (3):
  - Fundacion Hospital Infantil, Universitario De San Jose, Bogotá
  - Fundación Valle de Lili, Cali
  - Hospital Pablo Tobon Uribe, Medellín

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cohort 1 (Darifenacin 0.030 mg/kg/Day) | Cohort 2 (Darifenacin 0.0625 mg/kg/Day) | Cohort 3 (Darifenacin 0.125 mg/kg/Day)
Started | 12 | 14 | 9
Completed | 12 | 13 | 9
Not Completed | 0 | 1 | 0
Not completed — Protocol deviation | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety Population included all participants in the Full Analysis Set who took at least 1 dose of darifenacin.
Groups:
- Cohort 1 (Darifenacin 0.030 mg/kg/Day): Following a 7-day washout period, participants received darifenacin liquid oral suspension, 0.030 mg/kg/day dispensed per BID dosing, for 14 days.
- Total: Total of all reporting groups
Arm/Group | Cohort 1 (Darifenacin 0.030 mg/kg/Day) | Cohort 2 (Darifenacin 0.0625 mg/kg/Day) | Cohort 3 (Darifenacin 0.125 mg/kg/Day) | Total
Number analyzed (Participants) | 12 | 14 | 9 | 35
Age, Continuous [Mean (Standard Deviation); unit: years] | 9.2 (3.0) | 8.1 (3.2) | 7.3 (3.1) | 8.3 (3.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 8 | 5 | 16
  Male | 9 | 6 | 4 | 19

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Mean Maximum Bladder Capacity (MBC)
Description: MBC was defined as the volume of urine at which significant urinary leakage (i.e. leakage that prevents further volume increase) or significant discomfort/pain occurs, or a detrusor pressure at 40 centimeter (cm) H2O was reached.
Time Frame: Baseline (Day 0) to Day 14
Population: Per-protocol Population included all participants in the Safety Population who completed the study under treatment without major protocol deviation.
Measure: Mean (Standard Deviation); unit: milliliter (mL)
Arm/Group | Cohort 1 (Darifenacin 0.030 mg/kg/Day) | Cohort 2 (Darifenacin 0.0625 mg/kg/Day) | Cohort 3 (Darifenacin 0.125 mg/kg/Day)
Number analyzed (Participants) | 10 | 11 | 9
milliliter (mL)
  Baseline | 180.21 (126.88) | 142.18 (104.49) | 165.89 (123.74)
  Change From Baseline to Day 14 | -36.58 (93.59) | -14.64 (48.40) | 19.33 (76.12)

2. Secondary Outcome: Change From Baseline in Mean Volume at First Contraction
Description: Average volume of urine collected by catheterization at first contraction.
Time Frame: Baseline (Day 0) to Day 14
Population: Per-protocol Population included all participants in the Safety Population who completed the study under treatment without major protocol deviation. Number analyzed is the number of participants with available data at the given time point.
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Cohort 1 (Darifenacin 0.030 mg/kg/Day) | Cohort 2 (Darifenacin 0.0625 mg/kg/Day) | Cohort 3 (Darifenacin 0.125 mg/kg/Day)
Number analyzed (Participants) | 9 | 11 | 8
mL
  Baseline | 85.09 (71.65) | 56.91 (64.04) | 63.94 (51.38)
  Change From Baseline to Day 14 | -2.17 (62.79) | 14.00 (86.43) | 22.13 (85.53)

3. Secondary Outcome: Change From Baseline in Detrusor Pressure at First Contraction
Time Frame: Baseline (Day 0) to Day 14
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: cm H2O
Arm/Group | Cohort 1 (Darifenacin 0.030 mg/kg/Day) | Cohort 2 (Darifenacin 0.0625 mg/kg/Day) | Cohort 3 (Darifenacin 0.125 mg/kg/Day)
Number analyzed (Participants) | 9 | 11 | 8
cm H2O
  Baseline | 32.71 (43.35) | 16.36 (10.62) | 23.56 (19.25)
  Change From Baseline to Day 14 | -0.30 (13.85) | 0.36 (17.63) | 0.38 (16.86)

4. Secondary Outcome: Change From Baseline in Mean Volume at First Detectable Leakage
Description: Average volume of urine collected by catheterization at first detectable leakage.
Time Frame: Baseline (Day 0) to Day 14
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Cohort 1 (Darifenacin 0.030 mg/kg/Day) | Cohort 2 (Darifenacin 0.0625 mg/kg/Day) | Cohort 3 (Darifenacin 0.125 mg/kg/Day)
Number analyzed (Participants) | 8 | 10 | 5
mL
  Baseline | 151.25 (93.37) | 107.50 (117.50) | 113.70 (70.26)
  Change From Baseline to Day 14 | 26.40 (48.37) | -29.50 (67.40) | -31.40 (96.26)

5. Secondary Outcome: Change From Baseline in Mean Volume at 10, 20, 30, and 40 cm H2O Detrusor Pressure
Time Frame: Baseline (Day 0) to Day 14
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Cohort 1 (Darifenacin 0.030 mg/kg/Day) | Cohort 2 (Darifenacin 0.0625 mg/kg/Day) | Cohort 3 (Darifenacin 0.125 mg/kg/Day)
Number analyzed (Participants) | 10 | 11 | 9
mL
  Baseline at 10 cm H2O: number analyzed (Participants) | 9 | 11 | 7
  Baseline at 10 cm H2O | 58.58 (48.60) | 59.55 (49.98) | 83.71 (89.32)
  Change from Baseline to Day 14 at 10 cm H2O: number analyzed (Participants) | 9 | 11 | 7
  Change from Baseline to Day 14 at 10 cm H2O | 13.48 (94.96) | 0.27 (46.06) | 23.14 (91.69)
  Baseline at 20 cm H2O: number analyzed (Participants) | 8 | 9 | 5
  Baseline at 20 cm H2O | 85.30 (73.75) | 83.00 (69.81) | 106.60 (66.77)
  Change from Baseline to Day 14 at 20 cm H2O: number analyzed (Participants) | 8 | 9 | 5
  Change from Baseline to Day 14 at 20 cm H2O | -14.28 (65.95) | -3.11 (48.41) | -14.80 (71.48)
  Baseline at 30 cm H2O: number analyzed (Participants) | 8 | 6 | 5
  Baseline at 30 cm H2O | 121.81 (84.56) | 118.17 (111.80) | 136.00 (98.77)
  Change from Baseline to Day 14 at 30 cm H2O: number analyzed (Participants) | 8 | 6 | 5
  Change from Baseline to Day 14 at 30 cm H2O | -9.09 (58.70) | -55.67 (101.26) | 19.40 (94.69)
  Baseline at 40 cm H2O: number analyzed (Participants) | 6 | 6 | 3
  Baseline at 40 cm H2O | 130.02 (92.57) | 137.50 (126.04) | 116.67 (90.64)
  Change from Baseline to Day 14 at 40 cm H2O: number analyzed (Participants) | 6 | 6 | 3
  Change from Baseline to Day 14 at 40 cm H2O | -42.30 (56.14) | -55.17 (106.36) | -89.67 (91.72)

6. Secondary Outcome: Change From Baseline in Mean Catheterization Volume
Description: Average volume of urine was collected by catheterization and was recorded in a bladder diary. Bladder volume was assessed by urodynamics. The bladder diary entries completed on any 2 consecutive days after completing wash-out and prior to the baseline urodynamic examination on Visit 2 was used to calculate the baseline (Day-1) i.e. Visit 2 values. Similarly, the bladder diary entries completed on any 2 consecutive days during the week prior to the final study visit on Day 14 i.e. Visit 4 was used to calculate the Visit 4 values. The positive change from baseline indicates improvement.
Time Frame: Baseline (Day -1) to 2 consecutive days during the week prior to final study Day 14
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Cohort 1 (Darifenacin 0.030 mg/kg/Day) | Cohort 2 (Darifenacin 0.0625 mg/kg/Day) | Cohort 3 (Darifenacin 0.125 mg/kg/Day)
Number analyzed (Participants) | 9 | 8 | 8
mL
  Baseline | 93.57 (64.18) | 65.98 (56.32) | 115.18 (71.64)
  Change From Baseline to Day 14 | 14.36 (44.68) | 5.36 (24.17) | -5.50 (30.03)

7. Secondary Outcome: Change From Baseline in Total Pad Weight In-between Catheterizations
Description: Urodynamic test was used to assess the total pad weight in-between catheterizations. The change in total pad weight in-between catheterizations was recorded in the bladder diary. The bladder diary entries completed on any 2 consecutive days after completing wash-out and prior to the baseline urodynamic examination on Visit 2 was used to calculate the baseline (Day-1) i.e. Visit 2 values. Similarly, the bladder diary entries completed on any 2 consecutive days during the week prior to the final study visit on Day 14 i.e. Visit 4 was used to calculate the Visit 4 values. The positive change from baseline indicates improvement.
Time Frame: Baseline (Day -1) to 2 consecutive days during the week prior to final study Day 14
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: milligram (mg)
Arm/Group | Cohort 1 (Darifenacin 0.030 mg/kg/Day) | Cohort 2 (Darifenacin 0.0625 mg/kg/Day) | Cohort 3 (Darifenacin 0.125 mg/kg/Day)
Number analyzed (Participants) | 7 | 8 | 8
milligram (mg)
  Baseline | 1428.157 (687.549) | 764.250 (469.197) | 690.875 (452.234)
  Change From Baseline to Day 14 | -274.786 (416.441) | 289.000 (440.619) | 38.125 (354.528)

8. Secondary Outcome: Change From Baseline in Mean Catheterization Volume at First Awakening
Description: The change in urine volume at first awakening catherization was recorded by the participant in a bladder diary. Bladder volume was assessed by urodynamics. The bladder diary entries completed on any 2 consecutive days after completing wash-out and prior to the baseline urodynamic examination on Visit 2 was used to calculate the baseline (Day-1) i.e. Visit 2 values. Similarly, the bladder diary entries completed on any 2 consecutive days during the week prior to the final study visit on Day 14 i.e. Visit 4 was used to calculate the Visit 4 values. The positive change from baseline indicates improvement.
Time Frame: Baseline (Day -1) to 2 consecutive days during the week prior to final study Day 14
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Cohort 1 (Darifenacin 0.030 mg/kg/Day) | Cohort 2 (Darifenacin 0.0625 mg/kg/Day) | Cohort 3 (Darifenacin 0.125 mg/kg/Day)
Number analyzed (Participants) | 9 | 8 | 8
mL
  Baseline | 99.67 (61.14) | 107.44 (104.58) | 129.06 (69.40)
  Change From Baseline to Day 14 | 47.94 (53.79) | 23.69 (128.66) | -7.75 (51.49)

ADVERSE EVENTS:
Time Frame: From first dose of study drug to 30 days after the last dose of study drug (Up to 55 days)
Description: Safety Population included all participants in the Full Analysis Set who took at least 1 dose of darifenacin.
Arm/Group | Cohort 1 (Darifenacin 0.030 mg/kg/Day) | Cohort 2 (Darifenacin 0.0625 mg/kg/Day) | Cohort 3 (Darifenacin 0.125 mg/kg/Day)
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/14 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/14 | 1/9
Other Adverse Events (participants affected / at risk) | 6/12 | 6/14 | 4/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 (Darifenacin 0.030 mg/kg/Day) (N=12) | Cohort 2 (Darifenacin 0.0625 mg/kg/Day) (N=14) | Cohort 3 (Darifenacin 0.125 mg/kg/Day) (N=9)
Urinary tract infection (Infections and infestations) | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 (Darifenacin 0.030 mg/kg/Day) (N=12) | Cohort 2 (Darifenacin 0.0625 mg/kg/Day) (N=14) | Cohort 3 (Darifenacin 0.125 mg/kg/Day) (N=9)
Vertigo (Ear and labyrinth disorders) | 0 | 2 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 2
Dry mouth (Gastrointestinal disorders) | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 0 | 1 | 0
Pyelonephritis (Infections and infestations) | 0 | 1 | 0
Urethral injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0
Body temperature increased (Investigations) | 0 | 1 | 0
Cardiac murmur (Investigations) | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 0
Headache (Nervous system disorders) | 3 | 0 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 1
Renal pain (Renal and urinary disorders) | 0 | 1 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.